CLINICAL TRIAL: NCT03631472
Title: A Feasibility Study: A Safety Evaluation of RheOx on Patients With Chronic Bronchitis in the United States
Brief Title: Gala Early Feasibility Study of RheOx
Acronym: Gala_EFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gala Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS003
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Chronic Bronchitis; Copd Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: Treatment with RheOx
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- RheOx Treatment (Experimental): RheOx Treatment (i.e., Bronchial Rheoplasty)
  Interventions: Device: RheOx

INTERVENTIONS:
Device: RheOx — RheOx is a device-based, energy delivery system that delivers energy to ablate soft tissue such as the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.
  Other Names: Bronchial Rheoplasty; Gala Airway Treatment System

SUMMARY:
An early feasibility study (EFS) to assess the safety and clinical utility of RheOx on patients with chronic bronchitis in the United States.

DETAILED DESCRIPTION:
RheOx is a device-based, energy delivery system that delivers energy for the ablation of soft tissue such as the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.

Two sessions of treatment will be delivered one month apart. The right lung is treated at the first treatment session and the left lung is treated at the second treatment session (approximately one month after the right side is treated). Treatment will be delivered by a respiratory physician (interventional pulmonologist) in a tertiary teaching hospital during a bronchoscopic procedure. The bronchoscopy will be delivered during general anesthesia. It is anticipated that the bronchoscopic procedure will last less than 60 minutes in total. Treatment will be deemed to have been delivered following the successful treatment during the two bronchoscopies.

Subjects will be required to submit tests during the study including three CT scans (lung), respiratory function tests, exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed with chronic bronchitis for a minimum of two years, where chronic bronchitis is defined clinically as chronic productive cough for three months in each of two successive years in a patient in whom other causes of productive cough have been excluded.
2. Subject responds to the first two questions of the CAT must sum to at least 7 points. If the sum of the first two CAT questions is 6 points and the subject's total CAT score is greater than 20 points, the subject may be enrolled.
3. Subject has preprocedure post-bronchodilator FEV1 of greater than or equal to 30% and less than or equal to 80% of predicted within three months of enrollment.
4. Subject has had 1 or more COPD exacerbations, defined as an acute worsening in respiratory symptoms that requires additional treatment, in the 12-months prior to enrollment.
5. Subject has a SGRQ score of greater than or equal to 25 and CAT score of greater than or equal to 10.
6. Subject has a cigarette smoking history of at least ten packs years.
7. Subject in the opinion of the site investigator is able to adhere to and undergo two bronchoscopies and has provided a signed informed consent.

Exclusion Criteria:

1. Subject has lower respiratory infection (e.g., common cold, pneumonia, MAI, tuberculosis) within the six weeks prior to the initial treatment bronchoscopy or mild or moderate COPD exacerbation (per GOLD guidelines) within 4 weeks of the procedure.
2. Subject is taking > 10 mg of prednisolone or prednisone per day.
3. Subject has an implantable cardioverter defibrillator or pacemaker.
4. Subject has a history of cardiac arrhythmia within past two years.
5. Subject has history of unresolved lung cancer in last 5 years.
6. Subject has bullous disease as defined by bullae exceeding 3 cm in diameter on HRCT.
7. Subject has pulmonary nodule or cavity rthat in the judgement of the investigator may require intervention during the course of the study.
8. Subject has prior lung surgery, such as lung transplant, LVRS, lung implant/prosthesis, metal stent, valves, coils, bullectomy, segmentectomy, or lobectomy. Pneumothorax without lung resection is acceptable. Pleural procedures without surgery are acceptable.
9. Subject has clinically significant cardiomyopathy.
10. Subject has severe bronchiectasis as outlined in the report of the CT scan of the chest by the interpreting radiologist or in the view of the PI, those findings bronchiectasis or any other significant second lung disease, are the main drivers of the patient's clinical symptoms.
11. Subject actively smoked (including tobacco, marijuana, e-cigarettes, vaping, etc.) within the last 6 months.
12. Subject has the inability to walk over 100 meters in 6 minutes.
13. Subject has clinically significant serious medical conditions, such as: congestive heart failure, angina or myocardial infarction in the past year, renal failure, liver disease cerebrovascular accident within the past 6 months, uncontrolled diabetes, uncontrolled hypertension or autoimmune disease.
14. Subject has uncontrolled GERD.
15. Subject has sever pulmonary hypertension.
16. Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines).
17. Subject is pregnant, nursing, or planning to get pregnant during study duration.
18. Subject has received chemotherapy within the past 6 months or is expected to receive chemotherapy during participation in this study.
19. Subject is or has been in another clinical investigational study within 6 weeks of baseline.
20. Subject on anticoagulation for cardiovascular indications and is unable to have anticoagulants (i.e., Aspirin, Plavix, Coumadin) withheld for at least seven days prior to bronchoscopy in the opinion of the Investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2024-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Alabama Lung Health Center, Birmingham, Alabama
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - MedStar Health, Baltimore, Maryland
  - Beth Israel Deaconess, Boston, Massachusetts
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krimsky WS, Mammarappallil JG, Kim V, Bannan B, Charbonnier JP, Hatton BA, Sciurba FC. Airway Mucus Plugging in Chronic Bronchitis and the Impact of Bronchial Rheoplasty. Chest. 2026 Jan;169(1):73-83. doi: 10.1016/j.chest.2025.06.022. Epub 2025 Jun 24. PMID 40571054
- [Derived] Sciurba FC, Dransfield MT, Kim V, Marchetti N, Comellas A, Hogarth DK, Majid A. Bronchial rheoplasty for chronic bronchitis: 2-year results from a US feasibility study with RheOx. BMJ Open Respir Res. 2023 Dec 26;10(1):e001710. doi: 10.1136/bmjresp-2023-001710. PMID 38151258

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RheOx Treatment
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RheOx Treatment
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21
FEV1 percentage of Predicted FEV1 [Mean (Standard Deviation); unit: percentage] | 53.3 (15.8)
FEV1/FVC [Mean (Standard Deviation); unit: ratio] | 51.2 (14.3)
CAT Total Score [Mean (Standard Deviation); unit: units on a scale] — The instrument is the COPD Assessment Test (CAT). This instrument contains 8 questions (subscales) each scored by the patient on a 0-5 categorical scale where higher scores indicate worse symptoms. The scores of the 8 questions are summed, providing a total score ranging from 0 to 40. The 8 questions pertain to cough, phlegm, chest tightness, exertion/breathlessness, activity impairment, confidence about leaving the home, sleep quality and energy level.
  units on a scale | 26.9 (4.9)
SGRQ Total Score [Mean (Standard Deviation); unit: units on a scale] — The instrument is the St. George's Respiratory Questionnaire (SGRQ). This instrument contains 50 questions organized into 2 parts (3 components). The 3 components are symptoms, activities and impact. Scoring includes dichotomous answers (true/false) and various Likert scales. A scoring algorithm is provided; scores range from 0 to 100, with higher scores indicating more limitations.
  units on a scale | 60.1 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Safety Through 12 Months: Rate of Serious Adverse Events
Description: Rate of serious adverse events of interest through 12 months. Events of interest are death, COPD exacerbation requiring hospitalization, pneumothrax within 2 days of procedure, pneumonia within 7 days of procedure, respiratory failure or arrhythmia requiring intervention.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RheOx Treatment
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: Clinical Utility: SGRQ Score at 6 Months
Description: The change from baseline to 6 months in St. George's Respiratory Questionnaire (SGRQ) total score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RheOx Treatment
Number analyzed (Participants) | 20
units on a scale | -13.3 (11.7)

3. Secondary Outcome: Clinical Utility: SGRQ Score at 12 Months
Description: The change from baseline to12 months in St. George's Respiratory Questionnaire (SGRQ) total score
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RheOx Treatment
Number analyzed (Participants) | 21
units on a scale | -16.6 (13.3)

4. Secondary Outcome: Clinical Utility: CAT Total Score at 6 Months
Description: The change from baseline to 6 months in COPD Assessment Test (CAT) total score
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RheOx Treatment
Number analyzed (Participants) | 20
units on a scale | -7.6 (5.1)

5. Secondary Outcome: Clinical Utility: CAT Total Score at 12 Months
Description: The change from baseline to 12 months in COPD Assessment Test (CAT) total score
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RheOx Treatment
Number analyzed (Participants) | 21
units on a scale | -9.0 (6.3)

6. Other Pre Specified Outcome: Hospitalization Rate
Description: The rate of hospitalizations (events/pt/year)
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2023-06

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RheOx Treatment
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RheOx Treatment (N=21)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hyponatremia (Blood and lymphatic system disorders) | 1 (1)
stress cardiomyopathy (Cardiac disorders) | 1 (1)
hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RheOx Treatment (N=21)
Chest pain (General disorders) | 3 (3) — these events occurred during the post-treatment recovery period
Gastroenteritis (Infections and infestations) | 2 (2) — these events occurred during the post-treatment recovery period
abnormal finding on CT scan (Investigations) | 2 (2) — these events occurred during the post-treatment recovery period
headache (Nervous system disorders) | 4 (4) — these events occurred during the post-treatment recovery period
urinary retention (Renal and urinary disorders) | 2 (2) — these events occurred during the post-treatment recovery period
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 11 (11)
cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) — these events occurred during the post-treatment recovery period
lung nodule (Respiratory, thoracic and mediastinal disorders) | 4 (4)
sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) — these events occurred during the post-treatment recovery period
wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) — these events occurred during the post-treatment recovery period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03631472/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03631472/SAP_001.pdf